CLINICAL TRIAL: NCT02001155
Title: Comparing the Effect of the Water Drinking Test on Intraocular Pressure in Patients With Prior Trabeculectomy or Tube Shunt Surgeries
Brief Title: Comparing the Effect of the Water Drinking Test on Intraocular Pressure
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jonathon Myers, Associate Professor, Ophthalmology; Director of Clinical Fellowship, Wills Eye
Other Study IDs: WEH - 10-989E
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Water drinking test; trabeculectomy; tube shunt
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trabeculectomy: Individuals in this group will have undergone a trabeculectomy for the treatment of glaucoma.
  Interventions: Procedure: Water Drinking Test
- Tube Shunt: Individuals in this group will have undergone a tube shunt for the treatment of glaucoma.
  Interventions: Procedure: Water Drinking Test

INTERVENTIONS:
Procedure: Water Drinking Test — The Water Drinking test has been identified as a reliable and safe tool to predict maximum intraocular pressure values during a diurnal tension curve and to assess the efficacy of surgical interventions. Participants are asked to drink 10 ml/kg water (or approximately 0.33 ounces of water for every 2.2 pounds of weight or about 2.5 cups for a 150 lb. individual) over 15 minutes. Intraocular pressure is assessed every 15 minutes for one hour.

SUMMARY:
A test that was common in the 1960's and was used to detect primary open angle glaucoma was the water drinking test (patients drank 1 quart of water to stress the fluid drainage mechanism of the eyes. Intraocular pressure was then measured over the next hour). Recently this test has been demonstrated as a predictor of peak eye pressure during the day. The purpose of this study is to compare the results of the water drinking test between eyes that have undergone trabeculectomy and eyes that have undergone tube shunt surgery.

ELIGIBILITY:
Inclusion Criteria:

* prior trabeculectomy or tube shunt for the treatment of glaucoma
* age 21-90 years

Exclusion Criteria:

* inability to give informed consent
* current ocular infection
* more than 1 prior trabeculectomy, or more than 1 prior tube shunt
* previous refractive surgery
* pregnant women
* heart failure
* renal failure or uncontrolled urine retention
* corneal abnormalities preventing reliable IOP measurement

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will have open angle glaucoma and have undergone either tube shunt surgery or trabeculectomy. All participants will be matched for range of recent intraocular pressure (average over the prior three visits of <12 mm Hg, 12 to <18 mm Hg, or >18 mm Hg), as well as number of medications (none, 1-2, 3 or more).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 1 hour
  IOP is assessed every 15 minutes for one hour after the water drinking test is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Myers, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript is currently under development.

REFERENCES:
- [Background] Waisbourd M, Savant SV, Sun Y, Martinez P, Myers JS. Water-drinking test in primary angle-closure suspect before and after laser peripheral iridotomy. Clin Exp Ophthalmol. 2016 Mar;44(2):89-94. doi: 10.1111/ceo.12639. Epub 2015 Nov 10. PMID 26332426